CLINICAL TRIAL: NCT03619395
Title: Strategies to Optimize the Control of Cardiovascular Risk Factors in Patients After an Acute Coronary Syndrome
Brief Title: Risc Optimisation- Acute cor5onary Syndrome
Acronym: RiskOp-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Sonia Ruiz Bustillo, MD, Parc de Salut Mar
Other Study IDs: ParcSM
Record Dates: First submitted 2018-06-26; First posted 2018-08-07 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Acute Coronary Syndrome; Ischemic Heart Disease
Keywords: Cardiovascular Secondary prevention; Cardiovascular risk factors control
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the percentage of patients that reach the objective levels of LDL cholesterol, glycosylated hemoglobin and blood pressure recommended by clinical guidelines after an acute coronary syndrome, following strategies of pharmacological optimization based on algorithms. The investigators hypothesize that the use of algorithms designed and protocolized within a cardiac rehabilitation program after an ACS to optimize pharmacological treatment is effective and safe to improve the control of risk factors in patients with high cardiovascular risk.

DETAILED DESCRIPTION:
Despite the evidence, lipid-lowering pharmacological intervention in secondary prevention remains insufficient. These data are also confirmed in a study conducted in our environment where of a total of 423 high-risk patients only 29% had an optimal control of LDL-C levels and 36% of glycated hemoglobin levels. A possible explanation is the so-called therapeutic inertia defined as the failure of physicians to initiate or intensify an indicated therapy. The inadequate treatment of the risks factors in the high-risk population increases morbidity and mortality, so it is very relevant to find strategies that improve adherence to clinical practice guidelines.

Prospective observational study of a patient population after ACS that will be compared with a historical cohort. All participants will give informed consent before initiating procedures within the cardiac rehabilitation program.

Primary outcome: To analyze the percentage of patients that reach the objective levels of LDL cholesterol and glycosylated hemoglobin recommended by clinical guidelines following pharmacological optimization protocols based on algorithms developed for this study. These results will be compared with the historical cohort of our hospital (usual practice) Secondary outcome: to analyze if the results of the intensive intervention during the first year are maintained in the long term (5 years)

Baseline clinical, analytical, echocardiographic, coronary anatomy and pharmacological therapy data will be collected. After six weeks of lipid-lowering treatment, a first analytical control will be carried out and, following the specific algorithm designed for this study, oral pharmacological treatment will be adapted if the LDL-C target level is not met. After any change in therapy, a new analytical control will be performed after 8 weeks. Diabetic patients will also undergo a baseline analytical study, if the glycosylated hemoglobin values are not in the range recommended by the clinical practice guidelines, pharmacological treatment optimization will be initiated following the algorithm designed for the study. After three months of treatment, a new control and optimization of the treatment will be carried out according to the protocol designed.

A follow-up will be carried out after 6, 12 months and 5 years

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized with a diagnosis of acute coronary syndrome who have signed informed consent

Exclusion Criteria:

* patients with disability or refusal to sign informed consent or who have comorbidities with a life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that reach the objective levels of LDL cholesterol and glycosylated hemoglobin recommended in the clinical guidelines | 12 months
  LDL cholesterol and glycosylated hemoglobin levels

SECONDARY OUTCOMES:
Percentage of patients that reach the objective levels of LDL cholesterol and glycosylated the long term. | 5 years
  LDL cholesterol and glycosylated hemoglobin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sonia Ruiz Bustillo, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 12 months of study completion
Access Criteria: Requestors will be required to sign a Data Access Agreement